CLINICAL TRIAL: NCT05176223
Title: Optimizing Outcomes of Patients With Advanced HCC Undergoing Immunotherapy Through Novel 68Ga PSMA PET Imaging
Brief Title: 68Ga PSMA PET Imaging for the Treatment of Advanced Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-007799; NCI-2021-12377 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-11-22; First posted 2022-01-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (68GA PSMA PET/CT) (Experimental): Patients undergo 68GA PSMA PET/CT scans at baseline, and after 3, 6, 9, and 12 cycles of standard of care immunotherapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 Gozetotide; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 68Ga PSMA PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 Gozetotide — Undergo 68Ga PSMA PET/CT
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo 68Ga PSMA PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests whether 68-Gallium prostate specific membrane antigen (68Ga-PSMA) positron emission tomography (PET) imaging can improve the diagnosis and management of liver cancer that has spread to other parts of the body (advanced). PSMA is a protein that appears in large amounts on the surface of liver cancer cells. The radioactive chemical compound (68Ga-PSMA) has been designed to circulate through the body and attach itself to the PSMA protein on liver cancer cells. A PET scan is then used to detect the location of the tumor cells. 68Ga-PSMA PET may improve upon the diagnosis and management of liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the performance of novel biomarkers derived from PSMA PET/computed tomography (CT) to measure response compared to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, in advanced hepatocellular carcinoma (HCC) patients treated with immunotherapy.

II. To identify precision imaging biomarkers that can predict response of HCC to novel immunotherapy.

OUTLINE:

Patients undergo 68GA PSMA PET/CT scans at baseline, and after 3, 6, 9, and 12 cycles of standard of care immunotherapy in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed-up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pathologically confirmed HCC not amenable to curative resection, transplantation or ablative therapies
* Have radiographically measurable disease by RECIST
* Eligible for atezolizumab/bevacizumab front line therapy
* Male or female with age greater than 18 years, with the capacity and willingness to provide written informed consent

Exclusion Criteria:

* Pregnant and/or breast-feeding patients. A negative pregnancy test within 48 hours of the PET scan
* Patients with higher than the weight/size limitations of PET/CT scanner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Time to treatment response | Up to 12 cycles of treatment or 36 weeks
  Defined as the time from study registration to complete response/partial response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and per PSMA positron emission tomography (PET)/computed tomography (CT).
Progression free survival (PFS) at 6 months | At 6 months
  Defined as the length of time during and after treatment that a patient lives with cancer without the disease worsening, per RECIST and PSMA PET/CT
Time to progression | Up to 3 years
  Defined as the time from study registration to disease progression per RECIST 1.1 and PSMA PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen H. Tran, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT05176223/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT05176223/ICF_001.pdf